CLINICAL TRIAL: NCT06421285
Title: Effect of Preoperative Exercise on the Prevention of Secondary Lymphedema in Breast Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jae Yong Jeon, MD, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-0255
Record Dates: First submitted 2024-05-10; First posted 2024-05-20 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Breast Neoplasms
Keywords: Preoperative Exercise; Lymphedema; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Lymphedema | interventions — Exercise; Resistance Training

STUDY DESIGN:
Intervention Model Description: * Intervention group
  * Control group
Who Masked: Participant
Masking Description: * Patients aged 20 or older and younger than 80 years old who were first diagnosed with breast cancer
  * Patients scheduled to undergo neoadjuvant chemotherapy before surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Individually tailored exercise consisting of aerobic, strength, and flexibility exercises is prescribed, self-exercise compliance monitoring through an application, and diet management education through nutritional counseling.
  Interventions: Behavioral: Aerobic exercise, Strength training, Flexibility exercise
- Control group (No Intervention): One session of flexibility exercise education, diet management education through nutritional counseling

INTERVENTIONS:
Behavioral: Aerobic exercise, Strength training, Flexibility exercise — Aerobic exercise: 30-40 minutes/time, 3-5 times a week, intensity of 4-6 points on the Rating of Perceived Exertion(RPE) 10-point scale(A simple conversation is possible during exercise, but the intensity is such that you feel out of breath) Strength training: 2-3 times a week, 3 sets of 10 repetitions per movement
  * Upper extremities: Biceps brachii, triceps brachii, deltoid, pectoralis muscle exercise
  * Lower extremities: gluteus maximus, hamstrings, quadriceps exercise Flexibility exercise: Stretching and mobility exercises reflecting post-surgery rehabilitation
  Arms: Intervention group

SUMMARY:
Research purpose: Lymphedema is a very common complication in breast cancer patients. However, since there is currently no curable treatment, it is important to prevent and reduce the severity of lymphedema. The purpose of this study is to evaluate whether preoperative exercise is effective in preventing lymphedema after surgery. For secondary outcome, the preventive effects of exercise on other upper extremity dysfunctions (eg. pectoralis tightness, Axillary web syndrome, Adhesive capsulitis), which are common in breast cancer patients, were assessed.

DETAILED DESCRIPTION:
Study subjects:

* Patients aged 20 or older who were first diagnosed with breast cancer
* Patients scheduled to undergo neoadjuvant chemotherapy before surgery Study design: Prospective randomized controlled comparative clinical study
* Intervention is performed for at least 3 months during the neoadjuvant chemotherapy period before surgery.
* Treatment group: Individually tailored exercise consisting of aerobic, strength, and flexibility exercises is prescribed, self-exercise compliance monitoring through an application, and diet management education through nutritional counseling.
* Control group: One session of flexibility exercise training, diet management education through nutritional counseling

Result variable:

* Primary outcome variable:

  1) Incidence and severity of postoperative lymphedema: bilateral upper limb volume, ICG lymphography
* Secondary outcome variables:

  1. Clinical information: Demographic, disease and treatment-related data
  2. Physical-related: height/weight/waist circumference measurement, body composition test, physical examination (axillary membrane evaluation)
  3. Upper extremity function (shortening of the pectoralis major muscle, adhesive capsulitis): evaluation of shoulder range of motion, upper extremity muscle strength/grip strength
  4. Quality of life assessment: European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30(EORTC QLQ-C30), European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Breast cancer module 23(EORTC QLQ-BR23)

Assessment Schedule:

* Initial treatment and evaluation: Immediately after breast cancer diagnosis
* Follow-up evaluation: Immediately after completion of exercise intervention (preoperatively), and at 1, 3, and 6 months postoperatively.

Number of study subjects:

* This study will be conducted as a preliminary study for future research, and will be conducted on a total of 60 patients (30 in the experimental group and 30 in the control group) with an allocation ratio between groups of 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 or older and younger than 80 who were first diagnosed with breast cancer
* Patients scheduled for surgery and starting neoadjuvant chemotherapy before surgery

Exclusion Criteria:

* Patients with medical contraindications to exercise intervention or pain or musculoskeletal conditions that may limit active exercise intervention

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Bilateral upper limb volume | Immediately, Preoperatively, 1 month, 3 months, 6 months.
  Using a tape measure, measure the circumference from the wrist to the armpit every 4cm, then apply the ΣCircumference2/π formula to calculate the volume of the upper limb.
ICG lymphography | Immediately, 1 month, 6 months.
  Indocyanine green (ICG) contrast agent is injected subcutaneously in the distal area, and lymph fluid flowing to the proximal area through collateral lymphatic vessels is checked with an infrared camera.

SECONDARY OUTCOMES:
Body composition | Immediately, 6 months.
  After attaching electrodes to both hands and feet using the Inbody S10 equipment, quantitatively evaluate body composition by measuring human body impedance using multiple frequencies.
Shoulder range of motion | Immediately, Preoperatively, 1 month, 3 months, 6 months.
  Measurements are made according to a standardized protocol using a goniometer.
Upper limb strength, grip strength | Immediately, 6 months
  Using a digital hand held dynamometer, the strength of elbow flexion and extension, shoulder abduction, and flexor extensor muscles was measured.
  Measure grip strength using a digital hand held dynamometer
EORTC QLQ-C30 | Immediately, 6 months
  Evaluate the patient's quality of life through the corresponding questionnaire
EORTC QLQ-BR23 | Immediately, 6 months
  Evaluate the patient's quality of life through the corresponding questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jaeyong Jeon, Principal Investigator — Asan Medical Center; Heejeong Kim, Study Chair — Asan Medical Center; Seungwoo Cha, Study Chair — Asan Medical Center; Chul Jung, Study Chair — Asan Medical Center; Hwayeong Cheon, Study Chair — Asan Medical Center; Junghwa Do, Study Chair — Asan Medical Center; Woojin Jeong, Study Chair — Asan Medical Center; Doyoung Kim, Study Chair — Asan Medical Center
Locations (1):
- Seoul Asan Medical Center, Seoul, Seoul Special City, South Korea

IPD SHARING:
Plan to Share IPD: No